CLINICAL TRIAL: NCT02357914
Title: Freehand Ultrasound to Evaluate Scapular Kinematics in People With Paraplegia
Acronym: FUS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yasin Dhaher, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: FUS_81377
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Spinal Cord Injuries; Shoulder Impingement Syndrome
Keywords: Ultrasound; Shoulder; Spinal Cord Injury; Fluoroscopy
MeSH Terms: conditions — Spinal Cord Injuries; Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with paraplegia: Individuals with a spinal cord injury below T1

SUMMARY:
Shoulder pain is very common in people with spinal cord injury (SCI). Persons with high-level paraplegia have higher chances to suffer shoulder pain and injury than those with lower-level paraplegia due to the shoulder muscle imbalance. As people with SCI overuse the shoulder during routine daily activities, the onset of pain or injury lead to increased healthcare expenses, limitation in activity, depression, decreased participation, and reduced quality of life. One of the main reasons of shoulder pain is believed to have a altered scapular movement. To clarify the mechanism of the shoulder pain and injury, comprehensive understanding of three-dimensional scapular kinematics is required. Ultrasound is a low-cost and non-invasive imaging system and has been used to diagnose the shoulder pain and injury in individuals with SCI. A freehand ultrasound (FUS) combining ultrasound with motion capture system to evaluate scapular movement was developed and presented favorable results in able-bodied population. The purpose of this study is to compare the FUS and widely used skin-based method against a radiographic based gold standard in people with paraplegia, and to elucidate the relationship among scapular movement and shoulder pain, pathology. This study will also allow us to gain more understanding of how level of injury influences the scapular behavior during functional activities. The investigators believe more severe shoulder pain and pathology will be associated with greater abnormal scapular movement. The investigators also believe that people with high-level paraplegia will have greater scapular abnormality than people with low-level paraplegia during arm elevation and weight relief raise tasks. By completing this study, the investigators will expect to deliver a reliable and valid tool to evaluate scapular movement and gain a better understanding how the altered scapular movement is related to shoulder pain and pathology. The investigators will also learn how the level of injury affects the scapular behavior during functional activities. The results of this study may help the shoulder pain management leading to the improvement in the quality of life of individuals with SCI.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: Compare the freehand ultrasound (FUS) and skin-based markers methods with a well-established and accurate dynamic biplanar fluoroscopy combined with model-based tracking techniques to evaluate scapular kinematics.

Hypothesis 1: Throughout the arm elevation and weight relief raise, FUS measurements will have lower standard error of measurement, greater intra-rater repeatability, and better agreement with biplanar fluoroscopy techniques than skin-based method for scapular tilting, upward rotation, and external rotation.

Aim 2: Establish the convergent validity of FUS and skin-based markers method by describing the relationship between scapular kinematics and established measures of shoulder pain and pathology.

Hypothesis 2: Individuals with paraplegia diagnosed with more severe shoulder pain and signs of shoulder pathology will have reduced scapular posterior tilt, upward rotation, and external rotation during arm elevation and weight relief raise tasks compared to those with less shoulder pain and pathology.

Aim 3: Characterize the effect of lesion level on scapular behavior during arm elevation and weight relief raise tasks.

Hypothesis 3: When compared to individuals with low-level paraplegia, individuals with high-level paraplegia will have decreased posterior tilt, upward rotation, and external rotation during arm elevation and weight relief raise tasks.

Study Procedure

* Human Subjects Ten individuals with paraplegia aged from 18 to 65 years old will be recruited for Aim 1, 2, and 3. An additional 30 individuals with paraplegia will be recruited for Aim 2 and 3. The participants will be dichotomized between high-level group (at T7 and above) and low-level group (below T7).[3] Inclusion Criteria include the level of your spinal cord injury is determined as paraplegia more than one year ago. Use the manual wheelchair as the primary means of mobility (>80% of mobility). Subjects do not have a history of fractures or dislocations in the shoulder from which they have not fully recovered and do not have an implant/pacemaker in the torso and dominant arm, Subjects with neurologic deficit in the arm will be excluded, as these would impact scapular kinematics. Subjects with a history of traumatic injury to the upper limb that has not fully recovered and those with syrinx or complex regional pain syndrome involving the arms will be excluded as this could also affect our measures but be unrelated to dynamic scapular movement. Subjects who have impaired cognition or difficulty reading the informed consent will also be excluded. Based on literature and our previous experience, we expect at least 50% of the SCI population to have shoulder pain. We will determine the prevalence of shoulder pain as subjects are recruited. Participants may be recruited through the research registry for the Center of Rehabilitation Outcomes Research or Clinical Neuroscience Research Registry at Rehabilitation Institute of Chicago.
* Methods and Procedures

General questionnaire Basic demographics including age, gender, height, weight will be recorded. We will also record disability type, lesion level, motor scores (using the International Standards for Neurological Classification), date of injury, and handedness.

Motion capture Participants will transfer to a customized chair equipped with an adjustable guide bar in the sagittal, coronal, and scapular plane. The chair is designed to ensure consistency in arm movement from rest to elevated positions. Height and depth-adjustable pads and adjustable straps will provide supports to isolate the scapular kinematics and minimize trunk movement. Participants will wear a slim-fit white tank top or remove their shirt to allow for placing the markers on the trunk and dominant arm. Marker placement, determined by the International Society of Biomechanics,[4] will include the following bony landmarks: C7, T8, anterior sternoclavicular (sternum), xyphoid, acromion, lateral epicondyle, medial epicondyle, and greater trochanter. These markers allow measurement of trunk and upper arm movement during trials. A custom designed orthogonal attachment with markers allows tracking of the US probe through space during scanning. A custom-made triangular triad, with three reflective markers, will be attached to the flat superior bony surface of the acromion process. For each subject, a static capture of all markers will be collected in the standard anatomical neutral position to create the reference trial between the triad coordinate system and scapular coordinate system determined by the markers placed on the acromial angle, root of the scapular spine, and inferior angle. After the static capture, the markers on the acromial angle, root of the scapular spine, and inferior angle will be removed. Triad attachment will remain on the acromion process during the dynamic trial. Movement of the subject and ultrasound probe will be collected using a motion capture system.

Freehand ultrasound technique One operator will perform all ultrasound scanning. Imaging will consist of scanning of the scapula. Ultrasound video files will be collected during the trial. Scapular scanning consists of positioning the ultrasound probe along the spine and medial border of the scapula. The ultrasound probe will be fully contacted and manually held on different points along the scapular spine and medial border during the dynamic trials. Ultrasound gel is applied to the skin overlaying the scapula and the probe is oriented to maintain visualization of the border of the scapula in the image.

Dynamic biplanar fluoroscopy and model based tracking technique Study will take place at the Northwestern Memorial Hospital (NMH) where equipped a number of Siemens/Philips bi-planar fluoroscopic imaging systems, managed by Dr. Ellen Kruk. The equipments include Siemens Artis Zee biplane, Siemens Neurostar biplane, Philips Allura FD20 fluoroscopic imaging systems located at interventional radiology. 64-sliced Siemens Definition or Sensation computer tomography (CT) scanners or Siemens 3T magnetic resonance imaging (MRI) scanner will also be utilized to obtain the bone models of humerus and scapula.

Procedures Ten participants will be tested for Aim 1, 2, and 3 in NMH and additional 30 participants will be tested for Aim 2 and 3 in Biodynamics and Muscle Fiber Laboratories at Rehabilitation Institute of Chicago. For dynamic trial, each participant will perform arm elevation (AE) and weight relief raise (WR) trials in a random order. For AE trial, subjects will be in their own chairs. Subjects will elevate the arm from neutral to 150° in the sagittal, coronal, and scapular plane (30° anterior to the frontal plane). Subjects will use their own wheelchair during data acquisition for the WR trial, which entails lifting and holding the buttocks off the seat with an elbow locked position.[5, 6] A metronome at a frequency of 0.3 Hz will guide AE and WR trials. Once the subjects are on pace with the metronome, the researcher will trigger the ultrasound and motion capture systems simultaneously. Subjects will be given a rest period after each trial to prevent fatigue. Three dynamic trials will be collected in each task. For testing Aim 1 in NMH, ten out of the 40 subjects will visit the department of interventional radiology at the NMH for the dual fluoroscopy testing and a CT scan. The dual fluoroscopic imaging system may track the shoulder joint while the subject performs arm elevation and weight relief push-up trials.

Arm elevation trials The participants may be in their own chair for performing the arm elevation protocols. A guide bar will be placed in the sagittal, coronal, and scapular plane. Prior to the start of the protocols, we will ask the participant to wear a slim-fit white tank top or remove their shirt to allow for placing the motion sensors on the skin of the participants' thorax, scapula, and upper arm. The participants will be asked to keep the dominant arm by the side. Bony points of the shoulder will be marked. The ultrasound probe will be used to sweep over the surface of the shoulder. The participants may be asked to stay in this position while up to three readings (ultrasound scans). The participants will be then asked to elevate the arm to a flexed position. Bony landmarks on the shoulder will be marked. The ultrasound probe will be used to sweep over the surface of the shoulder while the participants have risen and lowered the arm. The participants may also be asked to complete similar motions while holding a weight. The participants can stop at any time if they experience any pain. The participants will be provided rest periods to prevent fatigue. Video cameras or photo cameras may be used to record scapular movement and the experiment setup. The soft-tissue and bone surface around the glenohumeral joint and scapula will be monitored with ultrasound during movement. These trials will take up to 60 minutes to complete.

Weight relief push-up trials The participants will be asked to keep both arms straight while you push-up in your own chair. The participants may be asked to repeatedly hold the push-up position while up to three readings (ultrasound scans). The ultrasound probe will be used to sweep over the surface of the shoulder while performing the push-up. The participants can stop at any time if they experience any pain. The participants will be provided rest periods to prevent fatigue. These trials will take up to 60 minutes to complete.

The participants will have the optional to examine the scapular movement measured using bi-planar fluoroscopy ⎯ a dynamic X-ray imaging device. The participants' shoulder joint movement will be recorded during arm elevation and weight relief push-up. Before or after the bi-planar fluoroscopic imaging, a research staff will send the subjects to NMH Radiology for CT scan or Center for Translational Imaging for MRI scan. The CT/MRI scan will be used to construct the scapular and humeral models and provide the position and orientation of the bones. If feasible the same visit/day will include dual fluoroscopy performed at NMH. Otherwise a second visit will be arranged for the fluoroscopy. A qualified radiology staff from Department of Interventional Radiology will perform the dual fluoroscopy. This study will compare the in vivo scapular movement between the FUS and biplanar fluoroscopy. Entire protocol will last up to three hours. A urine pregnancy test will be done for woman subject before the fluoroscopy test.

Shoulder pain and pathology measures We will evaluate shoulder pain using Wheelchair Users Shoulder Pain Index (WUSPI): The WUSPI is a 15-item self-report instrument that measures shoulder pain intensity in wheelchair users during various functional activities of daily living, such as transfers, wheelchair mobility, dressing, overhead lifting, and sleeping. [7] Each item is scored using a 10 cm visual analog scale anchored at the ends with the descriptors of "no pain" and "worst pain ever experienced." Individual item scores are summed to arrive at a total index score. The WUSPI is valid and reliable - test-retest reliability of the total index score was 0.99 and Cronbach's alpha (internal consistency) was 0.98.[8] A standardized physical examination has been previously used in our study and consists of common clinical test such as palpation over the bicipital groove/biceps tendon, Neer impingement test, Hawkin's-Kennedy test, and O'Brien's test for the labrum and acromioclavicular joint.[9] For each item, the sign/symptom of pain is scored as either absent (0), equivocally present (1), or definitely present (2).[9] Items are summed to create a total score.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Have paraplegia as a result of a spinal cord injury morn than one year;
* Able to perform push-ups independently and raise the arm above the head;
* Self-propel a manual wheelchair as the primary means of mobility

Exclusion Criteria:

* Have history of fractures or dislocations in the shoulder, elbow, or wrist from which you have not fully recovered;
* Have upper limb pain as a result of a complex regional pain syndrome;
* Have a implant or pacemaker within the torso or upper arm;
* Pregnant female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with spinal cord injury and the lesion level below T1
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Scapulothoracic joint range of motion, maximum, and minimum position | Two hours
  Anterior/posterior tilting, protraction/retraction, lateral/medical rotation

SECONDARY OUTCOMES:
Shoulder pathology score | 15 minutes
  The total scores summed by the physical examination of the shoulder pathology
Wheelchair User's Shoulder Pain Index | 10 minutes
  Self-reported pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Sheng Lin, PhD, Principal Investigator — Dept. Physical Medicine and Rehabilitation, Northwestern University; Yasin Dhaher, PhD, Study Director — Dept. Physical Medicine and Rehabilitation, Northwestern University; Michael Boninger, MD, Study Director — Dept. Physical Medicine and Rehabilitation, University of Pittsburgh
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided